CLINICAL TRIAL: NCT01464788
Title: ARTSS-2: A Pilot, Phase 2b, Randomized, Multi-center Trial of Argatroban in Combination With Recombinant Tissue Plasminogen Activator for Acute Stroke
Brief Title: Randomized Controlled Trial of Argatroban With Tissue Plasminogen Activator (tPA) for Acute Stroke
Acronym: ARTSS-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted prematurely at 90 of 105 planned patients due to the beneficial results of embolectomy clinical trials.
Sponsor: Andrew D. Barreto, MD (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor-Investigator, Andrew D. Barreto, MD, Assistant Professor of Neurology, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-11-0464
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Ischemic Stroke
Keywords: stroke; Argatroban; thrombin-inhibition; thrombolysis; anticoagulation
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — argatroban; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose Argatroban + rt-PA (alteplase) (Experimental): 100 micrograms/kilogram bolus, followed by 1 microgram/kilogram/minute IV infusion for 48 hours
  and
  rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
  Interventions: Drug: Low Dose Argatroban; Drug: rt-PA (alteplase)
- High dose Argatroban + rt-PA (alteplase) (Experimental): 100 micrograms/kilogram bolus, followed by 3 micrograms/kilogram/minute IV infusion for 48 hours
  and
  rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
  Interventions: Drug: High Dose Argatroban; Drug: rt-PA (alteplase)
- rt-PA (alteplase) (Active Comparator): rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
  Interventions: Drug: rt-PA (alteplase)

INTERVENTIONS:
Drug: Low Dose Argatroban — 100 micrograms/kilogram bolus, followed by 1 microgram/kilogram/minute IV infusion for 48 hours and rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
  Other Names: Argatroban
  Arms: Low dose Argatroban + rt-PA (alteplase)
Drug: High Dose Argatroban — 100 micrograms/kilogram bolus, followed by 3 micrograms/kilogram/minute IV infusion for 48 hours and rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
  Other Names: Argatroban
  Arms: High dose Argatroban + rt-PA (alteplase)
Drug: rt-PA (alteplase) — rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour

SUMMARY:
Randomized controlled clinical trial to estimate overall treatment benefit (improvement in disability) among stroke patients treated with rt-PA who are randomized to also receive either low-dose Argatroban, high-dose Argatroban or neither.

DETAILED DESCRIPTION:
Recombinant tissue plasminogen activator (rt-PA), the only proven treatment for acute ischemic stroke, fails to reperfuse brain in most patients with large thrombi. In our Phase 2a low-dose safety study (n=65), the two drugs appeared safe when delivered concomitantly and recanalization rates were greater than historical controls. This study will provide evidence-based hypotheses and data needed to design a larger definitive trial.

The purpose of this trial is to estimate overall treatment benefit (improvement in disability) among stroke patients treated with rt-PA who are randomized to also receive either low-dose Argatroban, high-dose Argatroban or neither.

ELIGIBILITY:
Inclusion Criteria:

* Disabling Ischemic stroke symptoms with onset < 3 hours treated with IV rt-PA by local standards*.

  * or ≤ 4.5 hours according to local standard of care.
* NIHSS ≥ 10* or any NIHSS with an intracranial clot should be demonstrated on neurovascular imaging (TCD or CTA) in any one of the following areas: distal internal carotid artery (ICA) carotid artery (CA), middle cerebral artery (MCA - M1 or M2), posterior cerebral artery (PCA - P1 or P2), distal vertebral or basilar artery.
* TCD criteria: Thrombolysis in brain ischemia (TIBI) 0, 1, 2 or 3 - CT-Angiogram: thrombolysis in myocardial ischemia (TIMI) 0 or 1 * NIHSS ≥ 10, demonstration of clot on neuroimaging is not necessary (i.e., enrollment can proceed with non-contrast head CT alone), but if performed, a clot must be demonstrated.
* For those patients who will undergo repeat CT-Angiogram at 2-3 hours, estimated glomerular filtration rate (eGFR) must be ≥ 60 mL/min/1.73m2.
* Females of childbearing potential must have a negative serum pregnancy test (HCG) prior to the administration of trial medication.
* Signed (written) informed consent by the patient or the patient's legal representative and/or guardian.

Exclusion Criteria:

* Patients whom the treating physician is planning (or could plan) to treat with intra-arterial thrombolysis or other endovascular procedures (i.e., mechanical clot retrieval) aimed at recanalization.
* Evidence of intracranial hemorrhage (ICH) on baseline CT scan or diagnosis of a non-vascular cause of neurologic deficit.
* National institute health stroke scale (NIHSS) Level of Consciousness score (1a) ≥ 2.
* Pre-existing disability with mRS ≥ 2.
* CT scan findings of hypoattenuation of the x-ray signal (hypodensity) involving ≥ 1/3 of the MCA territory.
* Any evidence of clinically significant bleeding, or known coagulopathy.
* INR >1.5.
* Patients with an elevated activated partial thromboplastin time (aPTT) greater than the upper limit of normal
* Patients currently, or within the previous 24 hours, on an oral direct thrombin inhibitor (i.e., dabigatran).
* Heparin flush required for an IV line. Line flushes with saline only.
* Any history of intra-cranial hemorrhage, known arteriovenous -malformation or unsecured cerebral aneurysms.
* Significant bleeding episode [e.g. gastrointestinal (GI) or urinary tract] within the 3 weeks before study enrollment.
* Major surgery or serious trauma in last 2 weeks.
* Patients who have had an arterial puncture at a non-compressible site, biopsy of parenchymal organ, or lumbar puncture within the last 2 weeks.
* Previous stroke, myocardial infarction (MI), post myocardial infarction pericarditis, intracranial surgery, or significant head trauma within 3 months.
* Uncontrolled hypertension [Systolic blood pressure (SBP) > 185 mmHg or diastolic blood pressure (DBP) >110 mmHg] that does not respond to intravenous anti-hypertensive agents.
* Surgical intervention (any reason) anticipated within the next 48 hours.
* Known history of clinically significant hepatic dysfunction or liver disease - including a current history of alcohol abuse.
* Abnormal blood glucose <50 mg/dL (2.7 mmol/L).
* History of primary or metastatic brain tumor.
* Current platelet count < 100,000/mm3.
* Life expectancy < 3 months.
* Patient who, in the judgment of the investigator, needs to be on concomitant (i.e., during the Argatroban infusion) anticoagulants other than Argatroban, including any form of heparin, unfractionated heparin (UFH), low molecular weight heparin (LMWH), defibrinogenating agent, dextran, other direct thrombin inhibitors or thrombolytic agents, glycoprotein llb/llla (GPIIb/IIIa) inhibitor or warfarin.
* Participated in any investigational study within 30 days before the first dose of study medication.
* Known hypersensitivity to Argatroban or its agents.
* Additional exclusion criteria if patient presents between 3-4.5 hours:

  1. Age >80
  2. Currently taking oral anticoagulants (regardless of INR)
  3. A history of stroke and diabetes.
  4. NIHSS > 25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06-11 (Actual); Study Completion 2015-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Barreto, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Sugg RM, Pary JK, Uchino K, Baraniuk S, Shaltoni HM, Gonzales NR, Mikulik R, Garami Z, Shaw SG, Matherne DE, Moye LA, Alexandrov AV, Grotta JC. Argatroban tPA stroke study: study design and results in the first treated cohort. Arch Neurol. 2006 Aug;63(8):1057-62. doi: 10.1001/archneur.63.8.1057. PMID 16908730
- [Background] Barreto AD, Alexandrov AV, Lyden P, Lee J, Martin-Schild S, Shen L, Wu TC, Sisson A, Pandurengan R, Chen Z, Rahbar MH, Balucani C, Barlinn K, Sugg RM, Garami Z, Tsivgoulis G, Gonzales NR, Savitz SI, Mikulik R, Demchuk AM, Grotta JC. The argatroban and tissue-type plasminogen activator stroke study: final results of a pilot safety study. Stroke. 2012 Mar;43(3):770-5. doi: 10.1161/STROKEAHA.111.625574. Epub 2012 Jan 5. PMID 22223235
- [Derived] Barreto AD, Ford GA, Shen L, Pedroza C, Tyson J, Cai C, Rahbar MH, Grotta JC; ARTSS-2 Investigators. Randomized, Multicenter Trial of ARTSS-2 (Argatroban With Recombinant Tissue Plasminogen Activator for Acute Stroke). Stroke. 2017 Jun;48(6):1608-1616. doi: 10.1161/STROKEAHA.117.016720. Epub 2017 May 15. PMID 28507269
- See also: University of Texas Houston Stroke Team Website — https://med.uth.edu/neurology/specialty-programs/ut-stroke/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who have had an ischemic stroke and admitted to the Accident and Emergency Department or Acute Stroke Unit by their treating physician receive IV Recombinant tissue plasminogen activator as per standard treatment, provided they are able to be treated within 4.5 hours of the onset of their stroke symptoms.
Pre-assignment Details: Patients who met the inclusion criteria received a head CT scan prior to initiation of rt-PA and the Argatroban infusion. If available, patients also underwent intracranial vessel imaging performed before or immediately after IV-tPA bolus (but before Argatroban bolus). Patients could not be randomized until after the CTA demonstrated an occlusion.
Groups:
- Low-dose Argatroban + Rt-PA (Alteplase): 100 micrograms/kilogram bolus, followed by 1 micrograms/kilogram/minute IV infusion for 48 hours.
  and
  Intravenous rt-PA (alteplase) 0.9mg/kg (max dose 90mg); 10% bolus and remaining over 1 hour.
- High Dose Argatroban + Rt-PA (Alteplase): Argatroban: 100 micrograms/kilogram bolus, followed by 3 micrograms/kilogram/minute IV infusion for 48 hours.
  and
  Intravenous rt-PA (alteplase) 0.9mg/kg (max dose 90mg); 10% bolus and remaining over 1 hour.
- Rt-PA (Alteplase) Only: Intravenous rt-PA (alteplase) 0.9mg/kg (max dose 90mg); 10% bolus and remaining over 1 hour.
Period: Overall Study
Arm/Group | Low-dose Argatroban + Rt-PA (Alteplase) | High Dose Argatroban + Rt-PA (Alteplase) | Rt-PA (Alteplase) Only
Started | 30 | 31 | 29
Completed | 30 | 29 | 29
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Patient had hemorrhage after tPA started | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Argatroban + Rt-PA: 100 micrograms/kilogram bolus, followed by 1 micrograms/kilogram/minute IV infusion for 48 hours and rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
- High Dose Argatroban + Rt-PA: 100 micrograms/kilogram bolus, followed by 3 micrograms/kilogram/minute IV infusion for 48 hours and rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
- Total: Total of all reporting groups
Arm/Group | Low Dose Argatroban + Rt-PA | High Dose Argatroban + Rt-PA | Rt-PA (Alteplase) | Total
Number analyzed (Participants) | 30 | 31 | 29 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 13 | 37
  >=65 years | 19 | 18 | 16 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (15.1) | 67.1 (13.4) | 68.9 (15.4) | 68.9 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 12 | 40
  Male | 17 | 16 | 17 | 50
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 21 | 65
  United Kingdom | 8 | 9 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 0 or 1 on Modified Rankin Scale
Description: Excellent functional outcome as measured by the number of patients with a 0 or 1 on the modified Rankin Scale (mRS) at day 90 as assessed by study personnel blinded to treatment.
Time Frame: 90 days
Population: One patient in the high dose group did not receive Argatroban and another in the high dose group was lost to follow up; however, an intention-to-treat analysis was used and all 31 enrolled patients were included.
Measure: Number; unit: participants
Arm/Group | Low Dose Argatroban + Rt-PA | High Dose Argatroban + Rt-PA | Rt-PA (Alteplase)
Number analyzed (Participants) | 30 | 31 | 29
participants | 9 | 10 | 6

2. Primary Outcome: Number of Participants With Symptomatic Intracranial Hemorrhage Within 48 Hours of tPA Administration
Description: Symptomatic intracranial hemorrhage (sICH) is defined as any evidence of bleeding on CT scan that in the opinion of the treating physician and/or an independent safety monitor is associated with a clinically significant neurological worsening. A four or more point increase in the NIHSS score from baseline (or last score obtained prior to blood found on CT scan) to subsequent CT scan at the time of potential worsening can be used as a guide by the clinical investigator or safety monitor for what represents a significant worsening in neurologic status but sICH can include any worsening deemed significant by the clinical investigator or independent safety monitor.
Time Frame: 48-hours
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Low Dose Argatroban + Rt-PA (Alteplase): 100 micrograms/kilogram bolus, followed by 1 micrograms/kilogram/minute IV infusion for 48 hours and rt-PA (alteplase) 0.9mg/kg (max dose 90mg) - 10% bolus, then 90% over 1-hour
Arm/Group | Low Dose Argatroban + Rt-PA (Alteplase) | High Dose Argatroban + Rt-PA (Alteplase) | Rt-PA (Alteplase)
Number analyzed (Participants) | 30 | 31 | 29
participants | 4 | 2 | 3

ADVERSE EVENTS:
Time Frame: Baseline to day 90
Description: AE's regardless of whether thought to be associated with the study or IMP under investigation were graded by the investigator and recorded on the Electronic Case Report Form. An AE form was completed for any intracranial Hemorrhage (ICH). A hemorrhage was labeled as symptomatic by either the local principal investigator of the safety monitor.
Arm/Group | Low Dose Argatroban + Rt-PA | High Dose Argatroban + Rt-PA | Rt-PA (Alteplase)
All-Cause Mortality (participants affected / at risk) | 5/30 | 3/31 | 5/29
Serious Adverse Events (participants affected / at risk) | 15/30 | 15/31 | 14/29
Other Adverse Events (participants affected / at risk) | 27/30 | 25/31 | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Argatroban + Rt-PA (N=30) | High Dose Argatroban + Rt-PA (N=31) | Rt-PA (Alteplase) (N=29)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 3 (3)
Nervous system disorders (Nervous system disorders) | 11 (11) | 10 (10) | 9 (9) — includes: symptomatic intracranial hemorrhage, neurological worsening, cerebral edema/ brain herniation, seizures, etc.
Electrolyte imbalance (General disorders) | 5 (5) | 3 (3) | 5 (5)
Death (General disorders) | 5 (5) | 3 (3) | 5 (5)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Renal and Urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Infections and Infestations (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Argatroban + Rt-PA (N=30) | High Dose Argatroban + Rt-PA (N=31) | Rt-PA (Alteplase) (N=29)
Immune system disorders (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Dental (General disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 5 (5) | 7 (8) | 9 (9)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 0 (0) | 4 (4)
Electrolyte imbalance (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood - circulation system (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Hematologic (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 4 (5)
Nervous system disorders (Nervous system disorders) | 16 (18) | 7 (10) | 4 (5)
Ear, Nose and throat (ENT) (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (6) | 8 (9) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 9 (11) | 6 (8) | 4 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (5) | 3 (3)
Endocrine disorders (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (8) | 2 (2) | 3 (4)
Infections and infestations (Infections and infestations) | 7 (9) | 10 (12) | 6 (6)

LIMITATIONS AND CAVEATS:
Study limitations include the open-label design that was necessary due to prohibitive costs of placebo manufacture and sham aPTT tests. Given that vessel imaging was not mandatory, a meaningful analysis of early recanalization rates was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes